CLINICAL TRIAL: NCT03779243
Title: Melatonin Treatment for Sleep Disturbance in Orthopaedic Trauma Patients
Brief Title: Treatment for Sleep Disturbance in Orthopaedic Trauma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael J. Gardner, PROFESSOR OF ORTHOPAEDIC SURGERY AT THE STANFORD UNIVERSITY MEDICAL CENTER, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-48700
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Sleep Disturbance; Trauma
MeSH Terms: conditions — Parasomnias; Wounds and Injuries | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5mg Melatonin and Sleep Education (Experimental): Participants will take 5mg Melatonin nightly, 1 hour before bedtime and be provided educational materials to improve sleep hygiene. They will have study visits in clinic as part of standard-of-care at 6 weeks and 12 weeks. They will complete Pittsburgh Sleep Quality Index and SF-36 Quality of Life questionnaires at enrollment and at their clinic visits.
  Interventions: Dietary Supplement: Melatonin 5mg and Sleep Education
- Placebo Control (Placebo Comparator): Participants will be given placebo pills to be taken daily 1 hour before bedtime and are a "sleep aid". Participants will not receive any sleep education materials. They will have study visits in clinic as part of standard-of-care at 6 weeks and 12 weeks. They will complete Pittsburgh Sleep Quality Index and SF-36 Quality of Life questionnaires at enrollment and at their clinic visits.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin 5mg and Sleep Education — Melatonin 5mg daily and sleep education for 6 weeks following injury or surgery.
  Arms: 5mg Melatonin and Sleep Education
Other: Placebo — Daily placebo pills for 6 weeks following injury or surgery.
  Arms: Placebo Control

SUMMARY:
The purpose of the study is to test the efficacy of sleep treatment in human patients following traumatic injury. Specifically, the study will determine if treatment consisting of melatonin and education related to sleep habits are effective in treating sleep disturbance and improving sleep quality in Orthopaedic trauma patients. We hope to learn if melatonin and sleep education effectively improve sleep following traumatic injury, and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* New patients visiting the Orthopaedic Trauma Clinic or undergoing orthopaedic surgery in Stanford Hospital following traumatic injury. Accidental traumatic fracture injuries that are operative and non-operative. Must be able to swallow tablets.

Exclusion Criteria:

* Documented head trauma. Cognitive impairments. Minors. Previously diagnosed sleep disorders. Sleep apnea. Enrolled in another study. Women who are pregnant or may become pregnant or are nursing. Hypertension. Diabetes. Endocrine, autoimmune, depressive, bleeding or seizure disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Mean Change in Pittsburgh Sleep Quality Index Score | Baseline, week 6, and week 12
  9-item self-rated questionnaire that assesses clinical sleep quality and disturbances. Global PSQI scores are sums of the component scores, and range from 0-21. Higher scores indicate worse sleep quality.

SECONDARY OUTCOMES:
36-Item Short Form Survey (SF-36) to measure quality of life | Baseline, week 6, and week 12
  36-item, patient-reported survey of patient health-related quality of life.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Mean Change from Baseline in Pain Scores on the Visual Analog Scale (VAS) | Baseline, week 6, and week 12
  VAS is scored on a continuum from 0-10 indicating "no pain" to "unbearable pain". Higher scores indicate more pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Gardner, MD, Principal Investigator — Stanford Department of Orthopaedic Surgery
Locations (1):
- Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swann MC, Batty M, Hu G, Mitchell T, Box H, Starr A. Sleep Disturbance in Orthopaedic Trauma Patients. J Orthop Trauma. 2018 Oct;32(10):500-504. doi: 10.1097/BOT.0000000000001276. PMID 30086043